CLINICAL TRIAL: NCT07216014
Title: Analysis of the Efficacy and Safety of Interleukin-23 Monoclonal Antibody in Inflammatory Bowel Disease: A Prospective Study
Brief Title: Interleukin-23 Monoclonal Antibody for Inflammatory Bowel Disease: Efficacy and Safety
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jiayin Yao, Associate Chief Physician, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-529
Record Dates: First submitted 2025-09-28; First posted 2025-10-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease and Ulcerative Colitis
Keywords: Interleukin 23
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Interleukin-23

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Inflammatory bowel disease (Experimental): Patients who have been diagnosed with moderate to severe CD or UC by the end of the study period
  Interventions: Drug: Interleukin 23; Device: Interleukin 23

INTERVENTIONS:
Drug: Interleukin 23 — After obtaining the patient's informed consent, the drug treatment mainly consisting of interleukin-23 monoclonal antibody was carried out. Basic information and medical history of the patients were collected, and the treatment process of the patients was followed up. The drug regimen was adjusted based on the physician's experience. Follow-up and disease assessment were conducted at 0, 4, 8, 16, 24, 48, and 54 weeks, respectively. Blood, stool, and tissue samples were collected at the corresponding follow-up time points for gastrointestinal endoscopy, imaging examinations, laboratory index tests, self-assessment of symptoms by the subjects, assessment of adverse reactions, and nutritional risk screening, etc. The efficacy and safety of IL-23 inhibitor treatment for CD or UC were comprehensively evaluated.
Device: Interleukin 23 — After obtaining the patient's informed consent, the drug treatment mainly consisting of interleukin-23 monoclonal antibody was carried out. Basic information and medical history of the patients were collected, and the treatment process of the patients was followed up. The drug regimen was adjusted based on the physician's experience. Follow-up and disease assessment were conducted at 0, 4, 8, 16, 24, 48, and 54 weeks, respectively. Blood, stool, and tissue samples were collected at the corresponding follow-up time points for gastrointestinal endoscopy, imaging examinations, laboratory index tests, self-assessment of symptoms by the subjects, assessment of adverse reactions, and nutritional risk screening, etc. The efficacy and safety of IL-23 inhibitor treatment for CD or UC were comprehensively evaluated.

SUMMARY:
Patients diagnosed with moderate to severe CD or UC by the end of the study period were selected. After obtaining informed consent, treatment with infliximab-based drugs was initiated. Basic patient information and medical history were collected. The treatment process was followed, and the drug treatment plan was adjusted based on physician experience. Follow-up and disease assessments were conducted at 0, 4, 8, 16, 24, 48, and 54 weeks. At corresponding follow-up time points, blood, stool, and tissue samples were collected for gastrointestinal endoscopy, imaging examinations, laboratory tests, symptom self-assessment by participants, adverse reaction assessment, and nutritional risk screening. The efficacy and safety of IL-23 inhibitor treatment for CD or UC were comprehensively evaluated.

After the study began, regular check-ups and evaluations were required when necessary or before medication administration. Venous blood samples were collected, or fecal collection boxes were provided for stool collection. When intestinal endoscopy was required for re-examination, one piece of normal and one piece of diseased intestinal mucosa tissue were collected each time. When surgery was required, two pieces of normal and two pieces of diseased intestinal mucosa tissue were collected each time. Sample collection does not affect the disease treatment and evaluation process. If any discomfort occurs during IL-23 inhibitor treatment, or if there are new changes in the condition or any unexpected situations, including hospitalization at other medical institutions, disability, etc., regardless of whether they are related to the study, participants should notify the investigator promptly to allow for judgment and appropriate medical treatment or advice to ensure safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 65 years at the baseline visit;
2. Patients diagnosed with CD and UC as per the Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (2023 · Guangzhou) and the Chinese Guidelines for the Diagnosis and Treatment of Ulcerative Colitis (2023 · Xi'an);
3. If the subject is a fertile female, a pregnancy test must be conducted at the baseline to rule out pregnancy. The entire trial process must follow the contraceptive recommendations of this project (see below); women without reproductive potential (defined as post-menopause or permanent surgical sterilization) do not need to undergo a pregnancy test at the baseline;
4. The subjects fully understand the purpose of the trial, and should have a basic understanding of the pharmacological effects of the trial drugs and the possible adverse reactions; in accordance with the spirit of the Helsinki Declaration, they voluntarily sign the informed consent form and comply with the requirements of this research protocol.

Exclusion Criteria:

1. Diagnosed with ischemic enteritis, infectious enteritis, radiation enteritis, NSAIDs-related enteritis, and other autoimmune enteropathies;
2. Unable to administer IL-23 inhibitors regularly by intravenous or subcutaneous injection;
3. Evidence of toxic megacolon was detected during screening;
4. Previously underwent small bowel resection, ileocecal resection, extensive colon resection, subtotal resection or total colon resection, rectal resection, ileostomy, colostomy;
5. Subjects who need surgery due to the condition or plan to undergo elective surgery during the study;
6. Complicated with severe liver and kidney dysfunction;
7. Complicated with active bacterial or viral infections, chronic infections;
8. Biologic agents are contraindicated such as active tuberculosis with positive chest X-ray or strongly positive tuberculin skin test, active tuberculosis within the past five years, myocardial infarction, heart failure or demyelinating neurological diseases;
9. Had severe opportunistic infections during screening, such as severe or recurrent herpes zoster, active cytomegalovirus infection, Pneumocystis jirovecii, Histoplasma capsulatum, etc. infections;
10. Have a history of gastrointestinal dysplasia, or any biopsy during endoscopic examination has revealed dysplasia, excluding completely resected low-grade dysplastic lesions; Patients with a known history of lymphoid tissue proliferative diseases (including lymphoma), or with signs and symptoms of lymphoid tissue proliferative diseases (such as lymphadenopathy and/or splenomegaly); Patients with current or past malignant tumors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Steroid-Free Clinical Remission | 12th to 16th week
  Clinical remission in CD is defined as a CDAI score of less than 150, achieved without the use of corticosteroids.Clinical remission in UC is defined as a modified Mayo score of 2 or less, with no individual subscore greater than 1, achieved without the use of corticosteroids.

SECONDARY OUTCOMES:
Clinical Response | 12th to 16th week;52th to 54th week
  CD:A decrease in CDAI score by 70 points or more from baseline is considered a clinical response. UC: A decrease in the Modified Mayo Score by at least 30% and an absolute reduction of at least 3 points from baseline signifies a clinical response.
Endoscopic Remission | 12th to 16th week;52th to 54th week
  An SES-CD score of 2 or less indicates endoscopic remission. UC: An MES of 1 or less is defined as endoscopic remission.
Mucosal Healing | 12th to 16th week;52th to 54th week
  CD:An SES-CD score of 0 is indicative of mucosal healing. UC:An MES of 0 represents mucosal healing.
Radiological Remission | 12th to 16th week;52th to 54th week
  Defined as the complete disappearance or minimization of intestinal inflammation on imaging studies, signifying no visible lesions, normalized wall thickness, absence of strictures or obstructions, and no new areas of disease. Radiographic remission is an important indicator of deep remission in disease treatment goals.
Radiological response | 12th to 16th week;52th to 54th week
  Typically defined as a significant reduction in the size of affected areas, decreased wall thickness, and decreased markers of inflammation observed through imaging methods such as MRI or CT scans. A radiographic response indicates a reduction in disease activity but may not represent complete disease remission.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khor B, Gardet A, Xavier RJ. Genetics and pathogenesis of inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):307-17. doi: 10.1038/nature10209. PMID 21677747
- [Background] Verstockt B, Salas A, Sands BE, Abraham C, Leibovitzh H, Neurath MF, Vande Casteele N; Alimentiv Translational Research Consortium (ATRC). IL-12 and IL-23 pathway inhibition in inflammatory bowel disease. Nat Rev Gastroenterol Hepatol. 2023 Jul;20(7):433-446. doi: 10.1038/s41575-023-00768-1. Epub 2023 Apr 17. PMID 37069321
- [Background] Hart A, Panaccione R, Steinwurz F, Danese S, Hisamatsu T, Cao Q, Ritter T, Seidler U, Olurinde M, Vetter ML, Yee J, Yang Z, Wang Y, Johanns J, Han C, Sahoo A, Terry NA, Sands BE, D'Haens G; GRAVITI Study Group. Efficacy and Safety of Guselkumab Subcutaneous Induction and Maintenance in Participants With Moderately to Severely Active Crohn's Disease: Results From the Phase 3 GRAVITI Study. Gastroenterology. 2025 Aug;169(2):308-325. doi: 10.1053/j.gastro.2025.02.033. Epub 2025 Mar 18. PMID 40113101